CLINICAL TRIAL: NCT05946746
Title: A Randomised, Double-blind, Placebo Controlled Study to Evaluate the Effect of PeptiStrong Supplementation in Conjunction with an Exercise Program to Enhance Muscle Strength in Young Subjects
Brief Title: The Effects of PeptiStrong and Exercise to Enhance Muscle Strength in Young Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PN23.002
Record Dates: First submitted 2023-06-07; First posted 2023-07-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Muscle Injury
Keywords: Muscle health; Muscle strength; Muscle fatigue; Muscle contraction; Physical endurance; Physical fitness; Musculoskeletal health; Body composition; Dietary supplements; Peptides

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PeptiStrong - fava bean hydrolysate preparation (Experimental): PeptiStrong 2.4g/day will be supplemented as 5 capsules (480mg each) taken with approx. 150mL water at breakfast once per day for 56 days
  Interventions: Dietary Supplement: PeptiStrong
- Silicated micro-crystalline cellulose (SMCC) (Placebo Comparator): The placebo 2.4g/day will be supplemented as 5 capsules taken with approx. 150mL water at breakfast once per day for 56 days
  Interventions: Dietary Supplement: Placebo SMCC silicated micro-crystalline cellulose

INTERVENTIONS:
Dietary Supplement: PeptiStrong — PeptiStrong is a protein hydrolysate derived from Vicia faba. It is a free-flowing powder, pale yellow in colour. For the purposes of the trial, PeptiStrong will be encapsulated in size '00' hydroxypropyl methylcellulose capsules.
  Arms: PeptiStrong - fava bean hydrolysate preparation
Dietary Supplement: Placebo SMCC silicated micro-crystalline cellulose — Placebo - SMCC silicated microcrystalline cellulose (INCI name: MCC, cellulose gel), For the purposes of the trial, SMCC will be encapsulated in size '00' hydropropyl methylcellulose.
  Arms: Silicated micro-crystalline cellulose (SMCC)

SUMMARY:
A randomised, double-blind, placebo controlled study to evaluate the effect of PeptiStrong supplementation in conjunction with an exercise program to enhance muscle strength and endurance in young male and female subjects.

DETAILED DESCRIPTION:
This study aims to further investigate the use of PeptiStrong as a sports supplement by evaluating its efficacy for improving muscle strength in healthy males and females. PeptiStrong will be supplemented as a single oral dose of 2.4g/day into the volunteers' diet for 56 days in conjunction with a predefined whole body exercise programme to be performed 3 times per week. The primary outcome will measure the difference in muscle strength as assessed by one-repetition maximum (1RM) using leg extension from baseline to Day 56 between PeptiStrong and placebo.

Secondary endpoints investigated during the trial will include changes in strength via the leg extension at Day 28 between PeptiStrong and Placebo, strength via bench press 1RM at Days 28 and 56, muscle endurance using 80% of baseline 1RM to failure via bench press and leg extension, number of repetitions on leg extension, muscle size measurements, muscle mass via DEXA scanning, arm, chest, thigh and waist circumference, safety and tolerability via adverse event reporting and vital sign recording. In addition to the measurements described above, volunteers will be asked to fill out a quality of life questionnaire for subjective endpoint analysis and also to record their food intake at predefined intervals during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males & females between 19 and 40 years of age
* BMI between 18.5 to 29.9 kg/m2, inclusive
* Females not of childbearing potential, defined as those who have undergone a sterilisation procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening, or, Individuals of child bearing potential must have a negative baseline urine pregnant test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control include:

Hormonal contraceptives including oral contraception, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant.

Double-barrier method Intrauterine devices Non-heterosexual lifestyle or agrees to use contraception if planning to change to heterosexual partner Vasectomy of partner at least 6 months prior to screening Abstinence and agrees to use contraception if planning on becoming sexually active

* Willing and be capable of performing the recommended physical training and exercise regimen (3 x/week) for the duration of the study, as determined by the QI
* Motivated to comply with exercise guidelines as assessed by the Self-motivation Questionnaire at screening
* Self-reported stable body weight for the past 3 months defined as not having gained or lost more than 5 kg of body weight throughout the 3 months prior to baseline as assessed by the QI.
* Agrees to refrain from taking NSAIDs and alcohol consumption for 24 and 48 hours, respectively, prior to each clinic visit
* Agrees to avoid vigorous exercise (e.g. running, swimming laps, tennis singles, uphill hiking, weight lifting) for 48 hours prior to the exercise challenge.
* Agrees to maintain current lifestyle habits as much as possible throughout the study depending on ability to maintain the following: diet and caloric intake, medications, supplements and sleep
* Willingness to complete questionnaires, records and diaries associated with the study and to complete all study assessments
* Provided voluntary, written, informed consent to participate in the study
* Healthy as determined by medical history, physical examination, ECG, and vital signs, as assessed by the QI

Exclusion Criteria:

* Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
* Allergy, sensitivity, or intolerance to the investigational product or placebo ingredients
* Has participated in structured resistance/power exercise training for >3 hours/week in the 6 months prior to baseline, as assessed by the QI
* Currently experiencing any medical condition (e.g., orthopedic injury, surgery, neuromuscular problems, musculoskeletal injury and/or disease) that may interfere with the ability to undergo physical strength testing during the study and/or ability to complete exercise guidelines as assessed by the QI
* Metal implants or other physical characteristics/limitations that may affect DEXA scan results, as assessed by the QI
* Participants who have followed a specific diet (e.g. ketogenic, paleo, high-protein, vegetarian etc) or have had a change of diet within 30 days of baseline as assessed by the QI
* Have a history of being diagnosed with phenylketonuria or another disease affecting amino acid metabolism (i.e., maple syrup urine disease, etc.)
* Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
* Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
* Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
* Current or history of significant diseases of the gastrointestinal tract, as assessed by the QI
* Current unstable significant psychiatric condition (e.g., clinical depression, eating disorders) and/or sleep disorders, as assessed by the QI
* Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
* Type I or Type II diabetes
* Current unstable diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
* Current use of any prescribed or over-the-counter medications and/or supplements that may affect muscle mass, muscle strength, or metabolism, as assessed by the QI
* Alcohol intake average ˃2 standard drinks per day as assessed by the QI
* Alcohol or drug abuse within the last 12 months
* Regular use of tobacco, vapes or nicotine products within 6 months of baseline and during the study period, as assessed by the QI
* Blood donation 30 days prior to screening, during the study, or a planned donation within 30 days of the last study appointment as assessed by the QI
* Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
* Individuals who are unable to give informed consent
* Any other condition, chronic disease, or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
randomised, double-blind, placebo controlled study to evaluate the effect of PeptiStrong in conjunction with an exercise program on muscle strength in young males and females. | 56 days supplementation
  A randomised, double-blind placebo controlled study to evaluate the effect of PeptiStrong, a fava bean derived protein hydrolysate versus placebo when supplemented in conjunction with an exercise program on muscle strength in young males and females. PeptiStrong or placebo will be orally administered once per day for 56 days. Whole body training programmes will be performed thrice weekly. The difference in muscle strength from a baseline measurement at day 0 (Visit 2) to day 56 (Visit 4) will be measured by a 1RM using a leg extension .

SECONDARY OUTCOMES:
To assess the effects of PeptStrong in conjunction with exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when consumed over a 56 day period in conjunction with an exercise program three times per week on strength via leg extension 1RM (V2-V3)
To assess the effects of PeptStrong in conjunction with exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when consumed over a 56 day period in conjunction with an exercise program three times per week on strength via bench press 1RM (V2-V4)
To assess the effects of PeptStrong in conjunction with exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when consumed over a 56 day period in conjunction with an exercise program three times per week on Muscle endurance using 80% of baseline 1RM to failure via leg and bench press (V2-4)
To assess the effects of PeptStrong in conjunction with exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when consumed over a 56 day period in conjunction with an exercise program three times per week on number of repetitions on leg extension (V2-4)
To assess the effects of PeptStrong in conjunction with exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when consumed over a 56 day period in conjunction with an exercise program three times per week on measurement of arm, chest, thigh and waist circumference (V2-4)
To assess the effects of PeptStrong in conjunction with exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when consumed over a 56 day period in conjunction with an exercise program three times per week on skeletal muscle mass and fat mass using DEXA (V1 and V4)

OTHER OUTCOMES:
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker interleukin-6 (IL-6).
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker lactate dehydrogenase (LDH).
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker C-reactive protein (CRP).
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker Creatine Kinase (CK)
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker tumour necrosis factor (TNFa)
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker acylcarnitine.
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on free fatty acids (FFA).
effect of PeptiStrong in conjunction with exercise on future exploratory endpoints including blood biomarkers of muscle homeostasis pre and post exercise | 56 days supplementation
  To evaluate the effect of a daily administration of PeptiStrong versus placebo, when supplemented over 56 days in conjunction with a whole body exercise program on blood biomarker nicotinamide adenine dinucleotide (NAD+).

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Science Inc. 275 Dundas Street, TD Tower A, Suite G02, London, Southwestern Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohan NM, Khaldi N, Keogh B, Franklyn Miller A. Randomised, double-blind, placebo-controlled study to evaluate the effect on human strength and endurance after resistance training and supplementation of Vicia faba protein hydrolysate compared with placebo. BMJ Nutr Prev Health. 2025 Mar 26;8(1):e001050. doi: 10.1136/bmjnph-2024-001050. eCollection 2025. PMID 40771513